CLINICAL TRIAL: NCT00001397
Title: Evaluation, Treatment and Training Protocol for Patients With Bone Marrow Failure States, Isolated or Multilineage Cytopenias, Metastatic Solid Tumors, or Hematologic Malignancies
Brief Title: Evaluation, Treatment, and Training for Patients With Blood Disorders
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 940010; 94-H-0010
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Hematologic Diseases
Keywords: Hematopoiesis; Thrombocytopenia; Anemia; Neutropenia; Dysplasia; Hematologic Malignancies
MeSH Terms: conditions — Hematologic Diseases; Thrombocytopenia; Anemia; Neutropenia; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: treated according to the guidelines of standard medical evaluation and care. No investigational treatments or procedures will be administered on this protocol.

SUMMARY:
This study is designed to allow the evaluation, follow-up, and medical care of patients with blood disorders not currently participating in a research study being conducted by the Hematology Branch of the National Heart, Lung and Blood Institute (NHLBI) or not being screened for participation in a study.

The purpose of this study is to allow investigation into the blood disorders of patients in order to teach, learn, and gather more information about diseases of the blood.

In addition, this study allows researchers the opportunity to evaluate patients referred to the Hematology Branch of the NHLBI with rare or undiagnosed diseases of the blood. This may be potentially beneficial to the patient and at the same time contribute to the development of new research ideas.

DETAILED DESCRIPTION:
This protocol is designed to allow the evaluation, follow up, and standard medical care of patients (and when appropriate, their stem cell donor) with bone marrow failure states, cytopenias, metastatic solid tumors, or hematologic malignancies not currently entered on an active NHLBI protocol or not being screened for an active NHLBI research protocol. Its purpose is to allow investigation into the hematologic problems of these patients for the primary purpose of teaching and furthering general hematologic knowledge. The ability to evaluate and treat patients with a wide variety of hematologic disease is critical to maintaining our accreditation as a hematology fellowship program and training our fellows to be competent hematologists, as well as for keeping all staff, including senior staff, up-to-date and familiar with the evaluation and treatment of patients with a wide spectrum of hematologic disease. It also allows the NHLBI investigators to evaluate patients referred with rare or as yet undiagnosed hematologic problems, both potentially benefiting the patient and stimulating new research directions for the NHLBI in the future. Periodic follow-up and treatment of patients previously entered on NHLBI protocols in order to monitor the long-term course of the underlying hematologic state and the consequences of experimental treatments is also required for fellowship training, and for maintenance of good referral relationships with patients and their physicians.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients (and when appropriate the patient's stem cell donor) may be entered on this protocol at the discretion of the Principal and/or Associate Investigators if :

An investigator decides that it is in the best interest of the patient/donor and the Branch for the patient to be enrolled in this protocol while awaiting a decision on eligibility for other protocols; or after enrollment on another protocol, or to allow careful evaluation of patients with unique or rare disorders of direct interest to the Branch; or with more common disorders for fellowship teaching purposes.

The patient or the patient's guardian is capable of informed consent and signs the consent form. The consent form will be signed by parents or guardians of patients under the age of 18.

Age greater than or equal to 2 and weight greater than 12 kg.

Ages: 2 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects age 2 or older and weighing greater than 12 kg, who meet entry criteria will be considered for participation on this protocol at the discretion of the Principal or Associate Investigator.
Sampling Method: Non-Probability Sample
Enrollment: 1452 (Actual)
Dates: Start 1993-11-08 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
To provide a mechanism for the evaluation, follow-up, and standard hematological care of patients by the Hematology Branch | 20 years
  To provide a mechanism for the evaluation, follow-up, and standard hematological care of patients by the Hematology Branch

CONTACTS AND LOCATIONS:
Overall Officials: Georg Aue, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Giudice V, Wu Z, Kajigaya S, Fernandez Ibanez MDP, Rios O, Cheung F, Ito S, Young NS. Circulating S100A8 and S100A9 protein levels in plasma of patients with acquired aplastic anemia and myelodysplastic syndromes. Cytokine. 2019 Jan;113:462-465. doi: 10.1016/j.cyto.2018.06.025. Epub 2018 Jun 27. PMID 29958797
- [Derived] Giudice V, Banaszak LG, Gutierrez-Rodrigues F, Kajigaya S, Panjwani R, Ibanez MDPF, Rios O, Bleck CK, Stempinski ES, Raffo DQ, Townsley DM, Young NS. Circulating exosomal microRNAs in acquired aplastic anemia and myelodysplastic syndromes. Haematologica. 2018 Jul;103(7):1150-1159. doi: 10.3324/haematol.2017.182824. Epub 2018 Apr 19. PMID 29674506
- [Derived] Giudice V, Feng X, Lin Z, Hu W, Zhang F, Qiao W, Ibanez MDPF, Rios O, Young NS. Deep sequencing and flow cytometric characterization of expanded effector memory CD8+CD57+ T cells frequently reveals T-cell receptor Vbeta oligoclonality and CDR3 homology in acquired aplastic anemia. Haematologica. 2018 May;103(5):759-769. doi: 10.3324/haematol.2017.176701. Epub 2018 Feb 1. PMID 29419434
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1994-H-0010.html